CLINICAL TRIAL: NCT05403632
Title: Influence of Mediterranean Dietary Habits on Pregnancy and Foetus Development: the Role of Epigenetics and Inflammation
Brief Title: Mediterranean Diet on Pregnancy and Foetus Development
Status: Recruiting | Type: Observational
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Licia Iacoviello, Professor, Neuromed IRCCS
Other Study IDs: DEP_012022
Record Dates: First submitted 2022-04-20; First posted 2022-06-03 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Pregnancy Outcomes; Fetal Development; Infant Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — venous blood samples, umbilical cord blood, saliva samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The Mediterranean-style diet has been associated with longevity, long-life wellbeing, lower risk of cardiovascular disease, cancer, obesity, and metabolic syndrome. Research is pointing to the benefits that MeD could have in pregnant. Pregnancy is a very complex period and recently, the attention has been focused on the possibility that healthy dietary patterns positively influence pregnancy and the development of organs in the offspring. The mechanisms through which MeD influences pregnancy and fetal growth may partly depend on its antinflammatory properties and possibly on changes in epigenetic mechanisms. Systemic inflammation might contribute to the association between maternal obesity and less favorable neurodevelopmental outcomes. The investigators aim to define how maternal adhesion to MeD may affect pregnancy and new-born development, hence representing a notable burden from a public health and social perspective. Main objective of this project is to build up a birth cohort suitable to investigate the role of maternal dietary habits on maternal and new-born health, with special focus on MeD and its possible mechanism of action through epigenetic and inflammation changes. To establish a mother/new-born cohort, collect detailed information on maternal dietary habits and set-up a biobank of biological samples to evaluate the association between dietary habits and pregnancy outcomes. The investigators will recruit 2000 pairs (mother, new-born) in different obstetrics departments. To investigate the association between maternal dietary habits, foetal growth and offspring development and possible mediation by the inflammation profile of the mother. To understand whether maternal dietary habits are associated with epigenetic changes in the offspring and if this process is driven by the inflammation profile of the mother. Venous blood samples will be obtained at the baseline and at each gestational period for ultrasound at 11-13 gestational weeks, 20-22 weeks and 30-32 weeks. Women will be followed-up with standard clinical and 2D ultrasound examinations at gestational weeks 11-13, 20-22 and 30-32 to evaluate the fetal growth. Offspring development will be assessed at 6, 12, 18, 24 months of age. After delivery, the investigators will collect umbilical cord blood and saliva samples from new-born using standard procedures. To understand if new-born epigenetics is associated with infant physical and neurocognitive development in the following 2 years.

DETAILED DESCRIPTION:
The Mediterranean diet (MeD) is an eating pattern typical of the Mediterranean basin and is characterized by a wide consumption of plant foods, cereals, legumes, fish, olive oil as main fat source, and moderate wine consumption.The Mediterranean-style diet has been associated with longevity, long-life wellbeing, reduced risk of cardiovascular disease, cancer, obesity, and metabolic syndrome. Research is now pointing to the benefits that adherence to a MeD could have in women, while pregnant. Pregnancy, indeed, is a very complex period where growth, development, and maturity take place. The future body, in addition to increasing its cellular mass, progressively acquires functional capabilities that would permit it to live and grow out of the mother's womb. The mechanisms through which MeD influences pregnancy and foetal growth may partly depend on its antinflammatory properties and possibly on changes in epigenetic mechanisms. Indeed, changes in epigenetic profiles could mediate links between specific intrauterine, early postnatal exposures and future mental health outcomes or immune status in offspring. Systemic inflammation might contribute to the observed association between maternal obesity and less favourable neurodevelopmental outcomes. Studies have demonstrated that DNA methylation is linked to an increased inflammatory response as well as increased risk of chronic disease. Still, there is a scarcity of studies analysing how maternal nutrition influences health and development outcomes in new-born, and how it alters potentially underlying molecular pathways. Here the investigators aim to better define how maternal adhesion to MeD may affect pregnancy and new-born development, which, in turn, affect the risk of disease during adulthood, hence representing a notable burden from a public health and social perspective. Should this hypothesis be confirmed, our findings may allow developing specific and targeted public health interventions, possibly personalized programs based on the peculiar characteristics shown by each pair (mother/new-born). To establish a mother/new-born cohort, collect detailed information on maternal dietary habits and set-up a biobank of biological samples to evaluate the association between dietary habits and pregnancy outcomes. The investigators will recruit 2000 pairs (mother, new-born) in different obstetrics departments of the Neuromed Clinical Research Network. To investigate the association between maternal dietary habits, foetal growth and offspring development and possible mediation by the inflammation profile of the mother. To understand whether maternal dietary habits (exposure) are associated with epigenetic changes in the offspring (outcome) and if this process is driven by the inflammation profile of the mother. To understand if new-born epigenetics is associated with infant physical and neurocognitive development in the following 2 years. The study population consists of pregnant women attending the Units of Obstetrics and Gynecology at Neuromed Clinical Research Network (Casa di Cura Villa del Sole, Salerno, Istituto Clinico mediterraneo, Agropoli (SA), Casa di Cura Villa dei Platani, Avellino e Clinica Mediterranea, Napoli). Inclusion into the study takes place during the first prenatal visit and within the first trimester of pregnancy, and involves women who express the willing to deliver at the aforementioned operating units. All recruited women will sign an informed consent to participate in the study and an informed consent for genetic studies. Each woman, as well as the father of the child, will sign the written consent to processing of personal and genetic data of their new-born. Exclusion criteria are: pregnancy with foetuses with known chromosomal or congenital malformation, history of inflammatory disease, use of immunosuppressant drugs, pre-existing diabetes or hypertension, conception by heterologous artificial insemination, malabsorptive bariatric surgery, eating disorders. Dietary habits will be assessed by one-year recall food frequency questionnaire at baseline and by a 24-hour dietary recall interview for a total of 7 days at three different time points at 11-13 gestational weeks, 20-22 weeks and 30-32 weeks. To monitor dietary habits during pregnancy in real time an Ecological Momentary Assessment will be used, based on a signal-contingent approach, so that women will be solicited to record their dietary consumption and other information at semifixed intervals. From both questionnaires, the investigators will calculate the Mediterranean Diet Score, the total Food Antioxidant Content (FAC) score, the Polyphenols Antioxidant Content (PAC) score, the inflammatory potential of the diet and extract micro and macronutrients daily intakes. Food processing will be evaluated by specific classification. Information on physiological and pathological history and other lifestyles (sleep characteristics, physical activity, smoking habits) will be obtained by validated questionnaires. Physical activity will be assessed using the Pregnancy Physical Activity Questionnaire (PPAQ). Maternal anthropometric assessment (height, weight, waist circumference and blood pressure) will be measured following standard techniques. Pre-pregnancy and post-partum weights will be evaluated according to World Health Organization classification criteria for body mass index (BMI). The rate of pregnancy weight gain will be assessed according to the Institute of Medicine BMI criteria for pregnant women. Gestational Diabetes Mellitus will be diagnosed according to the National Institute for Health and Care Excellence Diabetes in Pregnancy guidelines. Pregnancy and delivery complications will be obtained from the mother's medical records. The presence of the following obstetric and perinatal complications will be recorded: excessive weight gain, gestational diabetes, hypertension, eclampsia, spontaneous early and late abortion, spontaneous and iatrogenic preterm delivery or preterm premature rupture of membranes. Venous blood samples will be obtained at the baseline and at each gestational period in correspondence of the routinely visit for ultrasound at 11-13 gestational weeks, 20-22 weeks and 30-32 weeks. Blood will be processed and aliquots of serum, plasma ethylenediaminetetraacetic acid and buffy coats for DNA extraction will be obtained. Longitudinal association analysis will be performed using dietary mother habits before and during pregnancy as exposure and maternal health (weight gain, blood pressure, metabolic parameters) and pregnancy complications as outcomes. Seven measurements will be taken at each visit to measure foetal growth: Biparietal and Occipito-Frontal Diameters; Head Circumference; Transverse abdominal diameter; Anterio-posterior abdominal diameter; Abdominal Circumference and Femur Length. Intrauterine growth restriction will be defined as Delphi criteria. At birth the following parameters will be recorded in new-born to evaluate growth and development by trained nurses using standardized protocols: Apgar score, birthweight, length, upper arm length, upper thigh length, head circumference, abdominal circumference, skinfold thickness. Birthweight and gestational age at delivery will be used to categorize each neonate as small-for-gestational age, appropriate-for-gestational age, or large-for-gestational age, using a sex-specific reference. Gestational age will be confirmed through a first-trimester ultrasound. Preterm birth will be defined as births <37 weeks of gestation. The presence of the following perinatal complications will be recorded: neonatal acidosis, low Apgar score, perinatal mortality or presence of any major neonatal morbidity. Offspring development will be assessed at 6, 12, 18, 24 months of age for each baby. Mothers will report i) breastfeeding and weaning of the baby; ii) anthropometric assessments at each paediatric periodical check, iii) measures of cognitive development like age (days) at first word, age at object manipulation, level of social interactions of the baby and ability to imitate/respond to the language of adults, iv) sensory-related skills like ability to discriminate familial sounds and recognize familial faces (low/medium/high) and iv) any medical issue of the baby. Moreover, to evaluate neuro-cognitive development the investigators will use the Bayley Scales of Infant Development (BSID-II) score, the most widely used test of infant development. To understand whether maternal dietary habits (exposure) are associated with epigenetic changes in the new-born (outcome) and if this process is driven by the inflammation profile of the mother. To understand if new-born epigenetics is associated with infant physical and neurocognitive development in the following 2 years. After delivery, the investigators will collect umbilical cord blood and saliva samples from 2000 new-born using standard procedures. DNA will be extracted and after bisulfite conversion of DNA, Genome-wide methylation analysis will be performed. Analyses will be carried out through common statistical software like R and Statistical Analysis Software. Despite the difficulty of disentangling risk factors, the period of in utero development is one of the most critical windows during which adverse conditions and exposures may influence the growth and development of the foetus, as well as its postnatal developmental and behavioural outcomes. Prenatal and early postnatal periods are therefore crucial to identify critical windows of susceptibility. The investigators expect to find a direct association between dietary habits of the mother before and during pregnancy with maternal and new-born health, possibly mediated by inflammation pattern of the mother, that may result in changes of methylation patterns of the new-born, two secondary mechanisms involved in pregnancy and perinatal complications and foetus development.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women attending the Units of Obstetrics and Gynecology at Neuromed Clinical Research Network
* women within the first trimester of pregnancy
* women who express the willing to deliver at the aforementioned operating units

Exclusion Criteria:

* pregnancy with foetuses with known chromosomal or congenital malformation
* history of inflammatory disease
* use of immunosuppressant drugs
* pre-existing diabetes or hypertension
* conception by heterologous artificial insemination
* malabsorptive bariatric surgery
* eating disorders

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female
Study Population: The study population consists of pregnant women attending the Units of Obstetrics and Gynecology at Neuromed Clinical Research Network (Casa di Cura Villa del Sole, Salerno, Istituto Clinico mediterraneo, Agropoli (SA), Casa di Cura Villa dei Platani, Avellino e Clinica Mediterranea, Napoli). Inclusion into the study takes place during the first prenatal visit and within the first trimester of pregnancy, and involves women who express the willing to deliver at the aforementioned operating units. All recruited women will sign an informed consent to participate in the study and an informed consent for genetic studies. Each woman, as well as the father of the child, will sign the written consent to processing of personal and genetic data of their new-born.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
obstetric and perinatal complications | 9 months
  Pregnancy and delivery complications will be obtained from the mother's medical records. The presence of the following obstetric and perinatal complications will be recorded: excessive weight gain (kg), gestational diabetes (n,%), hypertension (n, %) , eclampsia (n, %), spontaneous early and late abortion (n, %), spontaneous and iatrogenic preterm delivery or preterm premature rupture of membranes (n, %).

SECONDARY OUTCOMES:
new-born growth and development | 9 months
  Seven measurements will be taken at each visit to measure foetal growth by using fetal ultrasound examination: Biparietal and Occipito-Frontal Diameters (in cm); Head Circumference (in cm); Transverse abdominal diameter (in cm); Anterio-posterior abdominal diameter (in cm); Abdominal Circumference (in cm) and Femur Length (in cm). Intrauterine growth restriction will be defined as Delphi criteria. At birth to evaluate growth and development by trained nurses using standardized protocols: Apgar score, birthweight (in kg), length (in cm), upper arm length (in cm), upper thigh length (in cm), head circumference (in cm), abdominal circumference (in cm). Birthweight (in kg) and gestational age (in weeks) at delivery will be used to categorize each neonate as small-for-gestational age, appropriate-for-gestational age, or large-for-gestational age, using a sex-specific reference. Gestational age (in weeks) will be confirmed through a first-trimester ultrasound examination.

OTHER OUTCOMES:
infant physical development | 24 months
  Offspring development will be assessed at 6, 12, 18, 24 months of age for each baby. Mothers will report i) breastfeeding and weaning of the baby by questionnaire; ii) anthropometric assessments at each paediatric periodical check, in particular height (cm) and weight (kg) will be measured; iii) any medical issue of the baby by questionnaire.
infant neurocognitive development | 24 months
  Mothers will report i) measures of cognitive development like age (days) at first word, age at object manipulation (days), level of social interactions of the baby and ability to imitate/respond to the language of adults ; ii) sensory-related skills like ability to discriminate familial sounds and recognize familial faces (low/medium/high).
  To evaluate neuro-cognitive development we will use the Bayley Scales of Infant Development (BSID-II) score, the most widely used test of infant development.

CONTACTS AND LOCATIONS:
Overall Officials: Licia Iacoviello, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- Istituto Clinico Mediterranea, Agropoli, SA, Italy